CLINICAL TRIAL: NCT02359994
Title: Prospective, Multicenter, Multidisciplinary, Controlled Clinical Investigation Evaluating the Safety and Efficacy of PerClot® Polysaccharide Hemostatic System
Acronym: CLOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Artivion Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PCT1101.011-C(02/15)
Record Dates: First submitted 2015-02-03; First posted 2015-02-10 (Estimated); Results first posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Blood Loss, Surgical
Keywords: hemostasis
MeSH Terms: conditions — Blood Loss, Surgical

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cardiac Surgery (Experimental): For cardiac procedures, the site of evaluation for satisfaction of intraoperative eligibility criteria will be any bleeding sites on the epicardium, along an aortic anastomotic suture line, or an aortotomy suture line. For example, the surgeon will perform dissection of adhesions per his or her conventional methods and bleeding will be controlled using means continually employed by the surgeon prior to surgical closure. Prior to application along an aortic anastomotic suture line or an aortotomy suture line, suture line gaps > 2mm and large needle holes > 2mm will be ligated prior to assessment of intraoperative eligibility criteria. Any bleeding site on the epicardium, or along an aortic anastomotic suture line, or an aortotomy suture line meeting the eligibility criteria will be evaluated for satisfaction. PerClot should be applied after drug reversal and the patient is taken off by-pass.
  Interventions: Device: PerClot Polysaccharide Hemostatic System; Device: Arista AH
- General Surgery (Experimental): For liver resection procedures, the resected liver surface will be the site of evaluation. The surgeon will perform resection of the diseased portion of the liver per his/her conventional methods. Bleeding from discrete vessels will be controlled using means conventionally employed by the surgeon. Vessels > 2mm in diameter will be ligated and any observed bile leaks controlled prior to assessment of intraoperative eligibility criteria.
  For total splenectomy procedures, the site of evaluation for satisfaction of the intraoperative eligibility criteria will be the retroperitoneal surface. The surgeon will perform the splenectomy per his/her conventional methods. Vessels > 2mm in diameter will be ligated prior to assessment of intraoperative eligibility criteria.
  Any bleeding site on the retroperitoneal surface/cavity or exposed parenchymal surface will be evaluated for satisfaction of the eligibility criteria.
  Interventions: Device: PerClot Polysaccharide Hemostatic System; Device: Arista AH
- Urologic Surgery (Experimental): For on-clamp partial nephrectomies, the site of evaluation will be the kidney bed surface. The surgeon will perform resection of the kidney per his or her conventional methods. Vessels > 2mm in diameter will be ligated and entries into the collecting system controlled prior to assessment of intraoperative eligibility criteria. Any bleeding site on the kidney bed will be evaluated for satisfaction of the eligibility criteria after clamp release.
  For radical nephrectomies, the site of evaluation will be the retroperitoneal surface/cavity. The surgeon will perform the procedure per his or her conventional methods. Vessels > 2mm in diameter will be ligated prior to assessment of intraoperative eligibility criteria. Any bleeding site on the retroperitoneal surface/cavity will be evaluated for satisfaction of the eligibility criteria.
  Interventions: Device: PerClot Polysaccharide Hemostatic System; Device: Arista AH

INTERVENTIONS:
Device: PerClot Polysaccharide Hemostatic System — During the intraoperative period, the subject will be evaluated for bleeding; only those who meet the intraoperative inclusion criterion will be enrolled into the study. After confirmation of the intraoperative eligibility criteria, the subject will be randomized to receive an adjunct application of PerClot. The prescribed hemostatic agent will be applied according to its Instructions for Use.
Device: Arista AH — During the intraoperative period, the subject will be evaluated for bleeding; only those who meet the intraoperative inclusion criterion will be enrolled into the study. After confirmation of the intraoperative eligibility criteria, the subject will be randomized to receive an adjunct application of the control device. The prescribed hemostatic agent will be applied according to its Instructions for Use.

SUMMARY:
This is a prospective, multicenter, multidisciplinary, controlled clinical investigation evaluating the safety and efficacy of PerClot in achieving intraoperative hemostasis compared to a similar marketed hemostatic device.

Three hundred and twenty four subjects across a maximum of 25 investigational sites undergoing open elective cardiac, general, or urological surgical procedures who meet the eligibility criteria will be intraoperatively randomized to receive no more than the entire contents of up to two 5 gram bellows of either the investigational device or a control hemostatic agent on a bleeding site, whose anatomic site is smaller than or equal to 25cm² and whose anatomic application site is smaller than or equal to 47cm², when bleeding is within the pre-defined bleeding severity range after any applicable conventional means for hemostasis are attempted as specified in the intraoperative procedures.

Each investigational site is expected to enroll approximately 13-40 subjects. All investigational sites will be located in the U.S. Follow-up will occur at hospital discharge and 6 weeks post-device application. For oncologic subjects, an additional follow up will occur at 24 months post device application.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative inclusion:

  * Subject is undergoing one of the following open elective cardiac, general, or urological surgical procedures: Cardiac procedure (Epicardium); Cardiac procedure (aortic anastomosis or aortotomy suture line); Liver resection; Total splenectomy; On-clamp partial nephrectomy; or Radical nephrectomy.
  * Subject is willing and able to give prior written informed consent for investigation participation; and
  * Subject is > 22 years of age.
* Intraoperative inclusion:

  * Subject is undergoing one of the following elective procedures: Cardiac procedure (Epicardium); Cardiac procedure (Aortic Anastomosis or Aortotomy suture line); Liver resection; Total splenectomy; On-clamp partial nephrectomy; or Radical nephrectomy.
  * Subject in whom all visible vessels or suture holes greater than or equal to 2mm in diameter have been ligated;
  * Subject in whom there is bleeding at the specified area for each surgical procedure after any applicable conventional means for hemostasis are attempted as specified by the intraoperative protocol;
  * Subject in whom the anatomic site is equal to or less than 25cm²;
  * Subject in whom the anatomic application site is equal to or less than 47cm²; and
  * Subject in whom the bleeding flux from the identified lesion is > 0.000040[g/(cm²•s)] and ≤0.013[g/(cm²•s)].

Exclusion Criteria:

* Preoperative Exclusion Criteria

  * Subject with known sensitivity to starch or starch-derived materials;
  * Subject who has a clinically significant coagulation disorder or disease, defined as a platelet count <100,000 per microliter, International Normalized Ratio >1.5, or a PTT more than 1.5 times outside the laboratory's normal reference range;
  * Subject who used corticosteroids (excluding inhalers, eye-drops, and dermatologic corticosteroids) within 6 weeks prior to surgery;
  * Subject who has been treated with an investigational product and has not completed the entire follow-up period for that investigational product;
  * Subject who is pregnant (as confirmed by pregnancy test), planning on becoming pregnant during the follow-up period, or actively breast-feeding; and
  * Subject with poor blood glucose control as per glycosylated hemoglobin > 9%.
* Intraoperative Exclusion Criteria

  * Subject undergoing a cardiac procedure in which there is no aortic anastomosis or aortotomy suture line to evaluate using the bleeding severity scale (i.e., not for treatment at the distal coronary artery bypass graft anastomosis);
  * Subject in whom any major intraoperative bleeding incidences during the surgical procedure occurred (i.e., subject with assignment of an American College of Surgeons Advanced Trauma Life Support Hemorrhage Class of II, III, or IV Hemorrhage);
  * Subject who has an active or potential infection at the surgical site, or whose surgical wound is defined as a wound classification of CO (Contaminated) or D (Dirty or Infected) based upon the Center for Disease Control and Prevention's wound classification system; and
  * Subject who has undergone platelet receptor GP IIb/IIIa antagonist therapy less than 48 hours prior to surgery.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2015-04; Primary Completion 2019-01-11 (Actual); Study Completion 2019-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael House, MD, Principal Investigator — Indiana University; Marc Moon, MD, Principal Investigator — Washington University School of Medicine; William Chapman, MD, Principal Investigator — Washington University School of Medicine; Ronald P Kaufman, MD, Principal Investigator — Albany Medical College; Edward Chen, MD, Principal Investigator — Emory University; Robin Kim, MD, Principal Investigator — University of Utah; Derek DuBay, MD, Principal Investigator — Medical University of South Carolina; Adam Yopp, MD, Principal Investigator — University of Texas Southwestern Medical Center; Michael Argenziano, MD, Principal Investigator — Columbia University; K. Scott Coffield, MD, Principal Investigator — Baylor Scott and White Research Institute; Sean Castellucci, DO, Principal Investigator — Manatee Medical Research Institute; Viraj Master, MD, Principal Investigator — Emory University; Kiran Turaga, MD, Principal Investigator — University of Chicago; Carlo B Ramirez, MD, Principal Investigator — Thomas Jefferson University; Keith B Allen, MD, Principal Investigator — St. Luke's Hospital; Elaine Tseng, MD, Principal Investigator — San Francisco VA; Michael Jessen, MD, Principal Investigator — University of Texas Southwestern Medical Center; Michael D'Angelica, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Jonathan Silberstein, MD, MPH, Principal Investigator — Tulane University School of Medicine; S.Chris Malaisrie, MD, Principal Investigator — Northwestern University; Charles St. Hill, MD, Principal Investigator — University of Nevada, Las Vegas; Douglas Scherr, MD, Principal Investigator — Weill Cornell Urology; Thomas Guzzo, MD, Principal Investigator — University of Pennsylvania; Aaron Milbank, MD, Principal Investigator — Minnesota Urology
Locations (1):
- Indiana University d/b/a/ Methodist Research Institute, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] House MG, Kim R, Tseng EE, Kaufman RP Jr, Moon MR, Yopp A, Master VA. Evaluating the safety and efficacy of a novel polysaccharide hemostatic system during surgery: A multicenter multispecialty prospective randomized controlled trial. Surg Open Sci. 2024 May 3;19:205-211. doi: 10.1016/j.sopen.2024.04.009. eCollection 2024 Jun. PMID 38800121

RESULTS

PARTICIPANT FLOW:
Groups:
- PerClot: Participants received up to two 5 gram bellows during study procedure.
- Arista: Active Control. Participants received up to two 5 gram bellows during study procedure.
Period: Overall Population Study
Arm/Group | PerClot | Arista
Started (Enrolled and Randomized) | 161 | 163
Treated | 160 | 162
Completed | 156 | 155
Not Completed | 5 | 8
Not completed — Adverse Event | 1 | 1
Not completed — Death | 1 | 5
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Canceled appointment and followed up with their primary care physician instead. | 1 | 0
Not completed — Remained in the long term care facility to which the subject was discharged. | 0 | 1
Period: Extended Oncology 24-Month Survival
Arm/Group | PerClot | Arista
Started (Oncology subjects continued to be followed for an extended survival assessment at 24 months post-randomization after the 6 week or 3 month evaluation period in the Overall Population Study.) | 85 (Oncology subjects in the PerClot group who completed either the 6 week or 3 month visit in the Overall Population Study.) | 93 (Oncology subjects in the Arista group who completed either the 6 week or 3 month visit in the Overall Population Study.)
Completed (Completed the 24-month visit.) | 65 | 72
Not Completed | 20 | 21
Not completed — Death | 19 | 21
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intention-to-Treat Population, which consists of all randomized subjects
Groups:
- PerClot: Participants received up to two 5 gram bellows during index procedure.
- Arista: Active Control. Participants received up to two 5 gram bellows during index procedure.
- Total: Total of all reporting groups
Arm/Group | PerClot | Arista | Total
Number analyzed (Participants) | 161 | 163 | 324
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age is unknown for one PerClot subject.
  years
    number analyzed (Participants) | 160 | 163 | 323
    (all) | 59.1 (13.76) | 59.2 (13.85) | 59.2 (13.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 65 | 121
  Male | 105 | 98 | 203
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 9 | 21
  Not Hispanic or Latino | 148 | 154 | 302
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 15 | 22
  White | 147 | 141 | 288
  More than one race | 2 | 5 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 161 | 163 | 324
Bleeding Severity Score [Count of Participants; unit: Participants] — The Bleeding Severity Score is a scale that measures the severity of a bleeding site and is based on the surface area of the bleed and the bleeding flux (rate of flow). It ranges from 0 to 5, with 0=No Bleeding, 1=Ooze, 2=Slight Bleeding, 3=Moderate Bleeding, 4=Severe Bleeding, and 5=Life-Threatening Bleeding.
  Participants
    0 | 0 | 0 | 0
    1 | 93 | 92 | 185
    2 | 68 | 71 | 139
    3 | 0 | 0 | 0
    4 | 0 | 0 | 0
    5 | 0 | 0 | 0
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Population: Systolic blood pressure is unknown for one PerClot subject.
  mmHg
    number analyzed (Participants) | 160 | 163 | 323
    (all) | 135.3 (18.48) | 131.4 (20.86) | 133.3 (19.78)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Population: Diastolic blood pressure is unknown for one PerClot subject.
  mmHg
    number analyzed (Participants) | 160 | 163 | 323
    (all) | 77.7 (11.98) | 74.9 (11.75) | 76.3 (19.78)
Height [Mean (Standard Deviation); unit: cm] | 173.3 (10.09) | 172.7 (9.69) | 173.0 (9.88)
Hematocrit [Mean (Standard Deviation); unit: percent blood volume] | 39.8 (4.40) | 39.7 (5.12) | 39.7 (4.77)
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 13.2 (1.57) | 13.1 (1.83) | 13.2 (1.70)
Platelet Count [Median (Full Range); unit: platelets*10^3/mcl] — Population: Platelet count is unknown for fifteen (15) PerClot subjects and ten (10) Arista subjects.
  platelets*10^3/mcl
    number analyzed (Participants) | 146 | 153 | 299
    (all) | 212 [101 to 682] | 227.0 [70 to 577] | 220.0 [70 to 682]
Temperature [Mean (Standard Deviation); unit: degrees Celsius] — Population: Temperature is unknown for one (1) PerClot subject and four (4) Arista subjects.
  degrees Celsius
    number analyzed (Participants) | 160 | 159 | 319
    (all) | 36.6 (0.42) | 36.6 (0.38) | 36.6 (0.40)
Therapeutic Area [Count of Participants; unit: Participants]
  Cardiac | 43 | 43 | 86
  General | 75 | 80 | 155
  Urology | 43 | 40 | 83
Type I Diabetes [Count of Participants; unit: Participants] | 2 | 1 | 3
Type II Diabetes [Count of Participants; unit: Participants] | 31 | 36 | 67
Weight [Mean (Standard Deviation); unit: kg] | 86.0 (19.90) | 87.0 (20.44) | 86.5 (20.15)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Achievement of Hemostasis at 7 Minutes
Description: The primary objective of this clinical investigation is to demonstrate non-inferiority in the achievement of hemostasis of the treated bleeding site at 7 minutes in participants receiving PerClot compared to those receiving a control hemostatic device. The primary endpoint is the percentage of participants achieving hemostasis of the treated lesion at 7 minutes in each treatment group.
Time Frame: 7 minutes following application
Population: As Treated Population, which consists of all subjects who were randomized and treated with either PerClot or Arista, with subjects analyzed according to the treatment group for the treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | PerClot | Arista
Number analyzed (Participants) | 160 | 162
Participants | 145 | 149
Statistical Analysis 1: Comparison: PerClot vs Arista; The primary efficacy hypothesis is that the percentage of participants achieving hemostasis of the treated bleeding site at 7 minutes in the overall PerClot group is non-inferior to the percentage of participants achieving hemostasis at 7 minutes in the Arista group, the active control; Test type: Non-Inferiority — Non-inferiority was assessed with a pre-specified non-inferiority margin of 10%, such that the endpoint is successfully met if the non-inferiority one-sided p-value is less than 0.025 or, equivalently, if the lower bound of a two-sided 95% confidence interval for the difference between PerClot and Arista hemostasis rates is greater than -10%; p = 0.005, Farrington-Manning score test; Difference in percentage of participants = -1.4, 95% CI 2-sided [-7.5 to 4.8] — Directionality for difference in the percentage of participants achieving endpoint: PerClot - Arista

2. Secondary Outcome: Number of Participants With Achievement of Hemostasis at 5 Minutes
Description: The secondary objective of this investigation is to compare the achievement of hemostasis of the treated bleeding site at 5 minutes for participants receiving PerClot compared to those receiving a control hemostatic device. The secondary endpoint is the percentage of participants achieving hemostasis of the treated bleeding site at 5 minutes in each treatment group.
Time Frame: 5 minutes following application
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PerClot | Arista
Number analyzed (Participants) | 160 | 162
Participants | 144 | 138
Statistical Analysis 1: Comparison: PerClot vs Arista; The secondary efficacy hypothesis is that the percentage of participants achieving hemostasis of the treated bleeding site at 5 minutes in the overall PerClot group is non-inferior to the percentage of participants achieving hemostasis at 5 minutes in the Arista group, the active control; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Farrington-Manning score test; Difference in Percentage of Participants = 4.8, 95% CI 2-sided [-2.4 to 12.0] — Directionality for difference in the percentage of participants achieving endpoint: PerClot - Arista

ADVERSE EVENTS:
Time Frame: Three (3)-months post-randomization for the first five subjects enrolled and 6-weeks post-randomization for subjects who enrolled thereafter.
Arm/Group | PerClot | Arista
All-Cause Mortality (participants affected / at risk) | 1/161 | 5/163
Serious Adverse Events (participants affected / at risk) | 44/161 | 44/163
Other Adverse Events (participants affected / at risk) | 89/161 | 78/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PerClot (N=161) | Arista (N=163)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 2 (2) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Pulseless Electrical Activity (Cardiac disorders) | 1 (3) | 0 (0)
Cardiogenic Shock (Cardiac disorders) | 0 (0) | 2 (2)
Heart Failure (Cardiac disorders) | 0 (0) | 2 (2)
Pericardial Tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Acute Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
Complete Heart Block (Cardiac disorders) | 1 (1) | 0 (0)
Aortic Regurgitation (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Asystole (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Flutter (Cardiac disorders) | 1 (1) | 0 (0)
Sick Sinus Syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Fibrillation With Rapid Ventricular Response (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileal Fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Perihepatic Fluid Collection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 3 (3)
Edema Limbs (General disorders) | 2 (2) | 0 (0)
Implant Site Fluid Collection (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 0 (0) | 2 (3)
Biloma (Hepatobiliary disorders) | 0 (0) | 1 (1)
Portal Vein Thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Skin Infection (Infections and infestations) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 1 (1)
Abdominal Infection (Infections and infestations) | 1 (1) | 1 (1)
Pelvic Infection (Infections and infestations) | 0 (0) | 1 (2)
Diabetic Foot Infection (Infections and infestations) | 0 (0) | 1 (1)
Hematoma Infection (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Biliary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Wound Dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Intraoperative Bleeding (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arteriovenous Fistula Site Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal Anastomotic Leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ureteric Anastomotic Leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic Spine Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Failure To Thrive (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Electrolyte Abnormality (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal Stromal Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intracranial Aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Infarct Cerebral (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Mania (Psychiatric disorders) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2) | 2 (2)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (5)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypoxic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diaphoresis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Thromboembolic Event (Vascular disorders) | 1 (1) | 4 (5)
Blood Loss Of (Nos) (Vascular disorders) | 0 (0) | 3 (3)
Hematoma (Vascular disorders) | 2 (2) | 0 (0)
Distributive Shock (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Uncontrolled Hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Bleeding (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PerClot (N=161) | Arista (N=163)
Anemia (Blood and lymphatic system disorders) | 19 (19) | 12 (12)
Leukocytosis (Blood and lymphatic system disorders) | 9 (9) | 12 (12)
Atrial Fibrillation (Cardiac disorders) | 10 (10) | 9 (9)
Constipation (Gastrointestinal disorders) | 16 (16) | 12 (13)
Abdominal Pain (Gastrointestinal disorders) | 14 (14) | 14 (14)
Nausea (Gastrointestinal disorders) | 13 (13) | 14 (14)
Fever (General disorders) | 12 (12) | 5 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 22 (22) | 23 (24)
Hyperglycemia (Metabolism and nutrition disorders) | 14 (14) | 12 (12)
Hypokalemia (Metabolism and nutrition disorders) | 11 (12) | 12 (12)
Acute Kidney Injury (Renal and urinary disorders) | 11 (11) | 10 (10)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 20 (20) | 18 (18)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 14 (15) | 10 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 9 (9)
Hypotension (Vascular disorders) | 12 (12) | 19 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators will postpone single-site publications until after publication or disclosure of data representative of the entire study (i.e., from all study sites).

DOCUMENTS (2):
  • Study Protocol (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT02359994/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/94/NCT02359994/SAP_001.pdf